CLINICAL TRIAL: NCT00118456
Title: A Phase I/II, Multicenter, Randomized Dose-Escalation Study of Oral AEE788 on Intermittent Dosing Schedules in Adult Patients With Advanced Cancer (Effective Amendment 5) Previously Entitled A Phase IA, Multicenter, Dose-Escalating Study of Oral AEE788 on a Continuous Daily Dosing Schedule in Adult Patients With Advanced Cancer
Brief Title: Study of Oral AEE788 in Adults With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEE788A2101
Record Dates: First submitted 2005-07-01; First posted 2005-07-11 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Cancer
Keywords: Advanced cancers; EGFR; Her2; VEGFR
MeSH Terms: conditions — Neoplasms | interventions — AEE 788

ARMS (2):
- 1 (Experimental): Continuous daily dosing
  Interventions: Drug: AEE788
- 2 (Experimental): Monday, Wednesday, Friday Dosing
  Interventions: Drug: AEE788

INTERVENTIONS:
Drug: AEE788

SUMMARY:
AEE788 is an orally active, reversible, small-molecule, multi-targeted kinase inhibitor with potent inhibitory activity against ErbB and VEGF receptor family of tyrosine kinases. It has an IC50 of less than 100 nM against p-EGFR, p-ErbB2, and p-KDR (VEGFR2). This study will assess the safety, pharmacokinetic (PK)/pharmacodynamic (PD) profiles and clinical activity of AEE788 in advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor
* Adequate hematologic, renal and hepatic function
* Age ≥ 18 years
* Karnofsky performance status score ≥ 70%
* Life expectancy ≥ 12 weeks

Exclusion Criteria:

* Active brain metastases
* Peripheral neuropathy > grade 2
* Diarrhea > grade 1
* Gastrointestinal (GI) dysfunction
* Compromised cardiac function
* Concurrent severe and/or uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2003-07; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose and dose-limiting toxicity of AEE788 | 4.5 years
Maximum-tolerated dose, safety and tolerability of AEE788 | 4.5 years

SECONDARY OUTCOMES:
Single dose and repeated dose pharmacokinetic profile of AEE788 | 4.5 years
Pharmacodynamic effects | 4.5 years
Changes in glucose metabolism/cell viability | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Yale Cancer Center, New Haven, Connecticut
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Institute of Drug Development/Cancer Therapy and Research Center, San Antonio, Texas